CLINICAL TRIAL: NCT06715683
Title: An Open-label, Randomized, 2-Part, 4-Period, 2-Sequence, Fully Replicated Crossover Study to Assess the Comparative Bioavailability of BMS-986278 To-be-marketed Formulation Compared to the Phase 3 Clinical Trial Formulation in Healthy Participants
Brief Title: A Study to Evaluate Comparative Bioavailability of BMS-986278 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IM027-1035
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics; Comparative Bioavailability; BMS-986278

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1, Sequence 1 (Experimental)
  Interventions: Drug: BMS-986278 Batched method, Dose A; Drug: BMS-986278 Batched method, Dose B
- Part 1, Sequence 2 (Experimental)
  Interventions: Drug: BMS-986278 Batched method, Dose A; Drug: BMS-986278 Batched method, Dose B
- Part 2, Sequence 1 (Experimental)
  Interventions: Drug: BMS-986278 Batched method, Dose A; Drug: BMS-986278 Continuous method
- Part 2, Sequence 2 (Experimental)
  Interventions: Drug: BMS-986278 Batched method, Dose A; Drug: BMS-986278 Continuous method

INTERVENTIONS:
Drug: BMS-986278 Batched method, Dose A — Specified dose on specified days
Drug: BMS-986278 Batched method, Dose B — Specified dose on specified days
  Arms: Part 1, Sequence 1; Part 1, Sequence 2
Drug: BMS-986278 Continuous method — Specified dose on specified days
  Arms: Part 2, Sequence 1; Part 2, Sequence 2

SUMMARY:
This is a trial to evaluate the comparative bioavailability of BMS-986278 to-be-marketed formulation compared to the phase 3 clinical trial formulation in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female individuals not of childbearing potential (INOCBP) and males, healthy as determined by medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and clinical laboratory assessment results as determined by the investigator.
* Body mass index (BMI) 18.0 to 32.0 kg/m2, inclusive.
* Body weight ≥ 50 kg for males and ≥ 45 kg for females.

Exclusion Criteria:

* Any significant acute or chronic medical illness as determined by the investigator.
* Current or recent (within 3 months of study intervention administration) gastrointestinal (GI) disease or other procedures (eg, bariatric procedures) that could affect drug absorption, distribution, metabolism, and excretion. Note: uncomplicated appendectomy and hernia repair are acceptable).
* Any major surgery within 4 weeks of study intervention administration on Day 1, including GI surgery (eg, cholecystectomy and any other GI surgery or perforation that could impact upon the absorption of study intervention [uncomplicated appendectomy and hernia repair are acceptable]).
* History of known risk of bleeding.
* Inability to tolerate oral medication.
* Individuals (only females) who are of childbearing potential.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-03-16 (Actual); Study Completion 2025-03-16 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Up to Day 24
Area Under the Concentration-time From Time Zero to Time Last Qualifiable Concentration (AUC(0-T)) | Up to Day 24
Area Under the Concentration-time From Time Zero Extrapolated to Infinite Time (AUC(INF)) | Up to Day 24

SECONDARY OUTCOMES:
Time of Maximum Observed Plasma Concentration (Tmax) | Up to Day 24
Terminal Phase Half-life (T-HALF) | Up to Day 24
Apparent Total Body Clearance (CLT/F) | Up to Day 24
Apparent Volume of Distribution (Vz/F) | Up to Day 24
Number of Participants With Adverse Events (AEs) | Up to 28 Days Post-discontinuation of Study Intervention
Number of Participants With Clinical Laboratory Abnormalities | Up to Day 25
Number of Participants With Vital Sign Abnormalities | Up to Day 25
Number of Participants With 12-Lead Electrocardiogram (ECG) Abnormalities | Up to Day 25

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Anaheim Clinical Trials (ACT), Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at:
  https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com